CLINICAL TRIAL: NCT07081373
Title: Efficacy of Repeat Dosing of Liposomal Bupivacaine on Postoperative Pain in Patients With Anal Fistula: A Multicenter, Randomized, Open-Label, Controlled Study
Brief Title: Study on Repeat Liposomal Bupivacaine for Post-Surgery Pain in Anal Fistula Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: The First Affiliated Hospital of Guizhou University of Traditional Chinese Medicine (Unknown); Maoming People's Hospital (Other); Dongguan Hospital of Traditional Chinese Medicine (Other); Xingyi People's Hospital (Unknown); Nanjing Hospital of C. M. (Unknown); People's Hospital of Xinjiang Uygur Autonomous Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-365
Record Dates: First submitted 2025-06-26; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Anal Fistula
Keywords: Anal fistula; Bupivacaine liposome; Postoperative pain; Repeat dosing
MeSH Terms: conditions — Rectal Fistula; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine Repeat Dosing Group (Experimental): A single dose of liposomal bupivacaine is administered at the conclusion of surgery without adjunctive analgesics, followed by a supplemental dose 72 hours postoperatively.
  Interventions: Drug: A single dose of liposomal bupivacaine is administered at the conclusion of surgery without adjunctive analgesics, followed by a supplemental dose 72 hours postoperatively.
- Liposomal Bupivacaine Single-Injection Group (No Intervention): A single dose of liposomal bupivacaine is administered at the conclusion of surgery without adjunctive analgesics.

INTERVENTIONS:
Drug: A single dose of liposomal bupivacaine is administered at the conclusion of surgery without adjunctive analgesics, followed by a supplemental dose 72 hours postoperatively. — At surgical closure, a single dose of undiluted liposomal bupivacaine (266 mg/20 mL) is administered without concurrent analgesics. The total 20 mL volume is divided into six equal aliquots (≈3.3 mL each) and infiltrated circumferentially around the incision using a 25-gauge or larger-bore needle. Injections target tissue layers above and below the fascia and within the subcutaneous plane, with frequent aspiration during administration to mitigate intravascular injection risk. Seventy-two hours postoperatively, a repeat dose of undiluted liposomal bupivacaine (266 mg/20 mL) is administered. Prior to infiltration, topical lidocaine cream is applied to the per-incisional skin for ≥20 minutes. The full 20 mL volume is then injected uniformly around the incision via circumferential needle advancement into pericicatricial tissues.
  Arms: Liposomal Bupivacaine Repeat Dosing Group

SUMMARY:
Anal Fistula refers to an abnormal infectious fistula tract between the anorectum and the perianal skin. The prevalence of anal fistula is approximately 8.6 cases per 100,000 individuals. It can occur at any age but is relatively more common in individuals aged 20-40 years, with a higher incidence in males than females.

Postoperative wound management is a critical component of the overall treatment for anal fistula patients. Regular postoperative wound care, such as dressing changes, can reduce recurrence rates, alleviate pain, and shorten hospitalization time. However, postoperative pain remains a major challenge in wound management following anal fistula surgery. This is largely attributed to inadequate current postoperative analgesic protocols.

With ongoing advancements in local anesthetics, liposomal bupivacaine has been applied for postoperative analgesia. It offers higher bioavailability and a prolonged half-life, providing up to 72 hours of sustained analgesic effect. Given the limitations of existing analgesic strategies for post-anal fistula surgery, developing more effective pain management approaches to reduce postoperative pain holds significant clinical importance.

Therefore, the investigators propose that a repeat-dosing strategy based on liposomal bupivacaine may provide superior postoperative pain control for anal fistula patients. To investigate this, the investigators designed a prospective, multicenter, randomized, open-label, controlled clinical trial. This study aims to evaluate the efficacy and safety of repeat-dose liposomal bupivacaine for postoperative analgesia following anal fistula surgery, thereby generating high-level evidence to support its clinical application in this context.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with anal fistula and scheduled to undergo anal fistula surgery;
* Aged between 18 and 60 years;
* ASA (American Society of Anesthesiologists) physical status class I-II;
* Patient provides written informed consent after understanding the study protocol.

Exclusion Criteria:

* Anal fistula caused by specific etiologies (e.g., tuberculosis);
* Concurrent acute perianal skin infection;
* Poorly controlled diabetes (HbA1c >9%);
* Chronic use of corticosteroids;
* History of radiotherapy or chemotherapy within the past 2 weeks;
* Pregnancy or lactation;
* Hypersensitivity to local anesthetics or any component of the investigational drug;
* History of substance abuse, illicit drug use, or alcohol abuse;
* Use or planned use of non-opioid/opioid analgesics within 12 hours before/during surgery;
* Concurrent treatment with anticonvulsants, MAO inhibitors, antidepressants, neuromuscular blockers, or anticholinergics within 2 weeks prior to surgery;
* Severe hepatic/renal impairment, cardiopulmonary dysfunction, coagulation disorders, or comorbidities contraindicating surgery;
* History of severe psychiatric disorders or cognitive impairment;
* Sensory disorders (e.g., hyperalgesia) or preexisting pain interfering with postoperative pain assessment;
* Contraindications to amide-type local anesthetics, opioids, or propofol;
* Participation in investigational drug trials within 90 days prior to enrollment;
* Other clinical/laboratory conditions deemed by investigators to preclude trial participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-07-16 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of the Numerical Rating Scale (NRS) for pain within 7 Days postoperatively (NRS-AUC0-168h) | 7 days postoperatively
  Numerical rating scale, a numerical rating scale where participants select a number from 0 to 10 based on their subjective pain experience. On this scale:
  0 represents no pain; 10 represents the most severe pain imaginable.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) for pain during wound dressing changes within 7 days postoperatively | 7 days postoperatively
  Numerical rating scale, a numerical rating scale where participants select a number from 0 to 10 based on their subjective pain experience. On this scale: 0 represents no pain; 10 represents the most severe pain imaginable.
Area Under the Curve (AUC) of the Numerical Rating Scale (NRS) for pain from 96 to 168 hours postoperatively (NRS-AUC96h-168h) | 96 to 168 hours postoperatively
Number of breakthrough pain episodes and corresponding Numerical Rating Scale (NRS) scores during episodes | 7 days postoperatively
  Numerical rating scale, a numerical rating scale where participants select a number from 0 to 10 based on their subjective pain experience. On this scale: 0 represents no pain; 10 represents the most severe pain imaginable.
Postoperative 7-day cumulative consumption of all analgesic drugs (calculated as morphine equivalents) | 7 days postoperatively
Postoperative 7-day cumulative consumption of rescue analgesic drugs (calculated as morphine equivalents) | 7 days postoperatively
Safety (including incidence of postoperative adverse events and serious adverse events): Adverse events and serious adverse events occurring within 14 days after medication were assessed | 14 days after medication were assessed
Postoperative heart rate monitoring: Heart rate at 24h, 48h, 72h, 96h, 120h, 144h, and 168h postoperatively. | At 24, 48, 72, 96, 120, 144, and 168 hours postoperatively.
Postoperative blood pressure monitoring: systolic blood pressure, and diastolic blood pressure at 24h, 48h, 72h, 96h, 120h, 144h, and 168h postoperatively. | At 24, 48, 72, 96, 120, 144, and 168 hours postoperatively.
SF-12 scores at preoperative, 1 week, 1 month, and 2 months postoperatively. | 1 week, 1 month, and 2 months postoperatively.
  The 12-Item Short Form Health Survey (SF-12) is a widely used concise instrument developed by the Medical Outcomes Study (MOS) to assess an individual's health-related quality of life (HRQoL), derived as an abbreviated version of the SF-36 scale. Overall scores range from 0 to 100, with higher scores representing better health status.
Preoperative, 14-day postoperative, and 1-month postoperative Wexner Incontinence Scores | Prior to surgery; 14 days after surgery; 1 month postoperatively.
  The Wexner Incontinence score, also termed the Cleveland Clinic Fecal Incontinence Severity Scoring System (CCIS) is a fecal incontinence score from 0-20; where 0 is perfect continence and 20 is complete incontinence.
Analgesia satisfaction: Postoperative analgesic satisfaction was assessed using a 5-point categorical scale at 24h, 96h, and 168h postoperatively. | At 24, 96, and 168 hours postoperatively.
  The Postoperative Analgesia Satisfaction Scale is an investigator-developed instrument where participants select a number from 0 to 4 based on their subjective experience, with higher scores representing greater satisfaction.
Wound healing rate within 8 weeks postoperatively. | 8 weeks postoperatively
  Wound Healing Rate: The wound area on postoperative day 1 is defined as the initial wound area. Measure the maximum length and perpendicular width of the wound to calculate the wound area.
  Formula: Wound Healing Rate = [(Initial Area - Current Area) / Initial Area] × 100%.
Wound healing time within 8 weeks postoperatively. | 8 weeks postoperatively
  Wound Healing Time: The duration from initial dressing change until complete wound epithelialization is achieved.
Wound Edema Score within 8 weeks postoperatively. | 8 weeks postoperatively
  Wound Edema Scoring Criteria:
  3 points: Severe edema with gross elevation beyond wound margins, requiring surgical intervention; 2 points: Significant edema extending beyond wound margins, managed with dressing changes;
  1 point: Mild localized edema; 0 points: No detectable edema.
Wound granulation tissue color score within 8 weeks postoperatively. | 8 weeks postoperatively.
  Granulation Tissue Color Scoring:
  1. point: Bright red;
  2. points: Pale red;
  3. points: Purple.
Whether the wound is infected within 8 weeks postoperatively. | 8 weeks postoperatively.
Whether the wound is bleeding within 8 weeks postoperatively. | 8 weeks postoperatively.
  Whether bleeding is present (none, oozing, active)

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT07081373/Prot_SAP_000.pdf